CLINICAL TRIAL: NCT04321473
Title: Web-based Registry on Left Main From the Euro Bifurcation Club (WE REMAIN EBC)
Brief Title: Registry on Left Main Coronary Artery Bifurcation Percutaneous Intervention
Acronym: WE REMAIN EBC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: G. d'Annunzio University (Other)
Collaborators: Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti (Other); Hospital Clínico Universitario de Valladolid (Other); VZW Cardiovascular Research Center Aalst (Other); Federico II University (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Clinica Mediterranea (Other); Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other); San Raffaele University Hospital, Italy (Other); Instituto Dante Pazzanese de Cardiologia (Other); University Medical Centre Maribor (Other); Clinica Di Montevergine (Other); Clinical Hospital Centre Zagreb (Other); Clinical Centre of Serbia (Other); Chiba University (Other); Université Paris-Sud (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Mount Sinai Hospital, New York (Other); Hospital Pablo Tobón Uribe (Other); Pauls Stradins Clinical University Hospital (Other); University Hospital Monastir, Tunis (Other)
Responsible Party: Principal Investigator, Marco Zimarino, MD, PhD, G. d'Annunzio University
Other Study IDs: WE_REMAIN_EBC_19
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Coronary Arteriosclerosis; Left Main Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PCI on left main — PCI on left main coronary stenosis

SUMMARY:
The slowly accruing evidence on the treatment of patients with left main coronary artery (LMCA) disease drove evolution in guidelines, that currently establish equivalent safety and efficacy for percutaneous coronary intervention (PCI) as compared to surgery, with a class of recommendation that is subjected to the extension and complexity of concomitant coronary artery disease, as assessed by the SYNTAX score.

The severity of LMCA disease, although extremely relevant due to the extent of the supplied myocardium, is often difficult to assess with traditional angiography, due to lack of appropriate angiographic views, absence of a true "reference" segment, interaction with the intubating catheter. Intravascular techniques with either imaging or functional assessment have been variously tested, although with a disturbing rate of discordant results; moreover, they are frequently underused for a number of reasons, including the additional time needed to assess both left anterior descending (LAD) and left circumflex (LCx) arteries, technical challenges, costs and the small risk associated with maneuvering such devices. Fractional flow reserve (FFR) measured from the coronary angiogram (FFRangio) alone recently documented a high diagnostic accuracy compared with pressure-wire derived FFR.

As for the anatomical localization, the majority of LMCA lesions occur at the bifurcation, where PCI results are less favourable. The distal LMCA differs from the other bifurcations in several characteristics: a) a notable mismatch between the LMCA and the left anterior descending (LAD) artery, hampering the selection of an adequately sized stent, b) the presence of a trifurcation, with a large ramus arising from LMCA in about 10% of cases, c) the presence of left or co-dominant circulation, with the LMCA supplying all or nearly all left ventricular myocardium in about 15% of cases.

Therefore, although the European Bifurcation Club (EBC) recommends a provisional side branch approach in most cases of distal LMCA disease, the threshold for placing a second stent in the side branch may be lower in lesions located on LM bifurcation compared with non-LMCA bifurcations. As for double stenting, the evidence is controversial and a consensus is lacking. Moreover, the optimal treatment of patients with LM trifurcations is still undefined.

The aim of this study is therefore to determine the optimal strategy for the treatment of LM bifurcated lesions.

DETAILED DESCRIPTION:
PCI access site and technique will be left at the operator's discretion, as well as antithrombotic management.

No limitation will be applied for the technique of PCI. As regards data collection and endpoints, Case Report Form (CRF) will be entered on a web-based platform, where study participants will be able to access and retrieve data at any time during study progress.

In-hospital outcomes will be recorded; all patients discharged alive will be followed up with a 30-day, 6-month, and 1-year telephone interview.

On a center-to-center voluntary basis, pre-PCI and post-PCI angiographic images (made blind regarding patients' identity) will be sent to a study angiographic core-lab for Quantitative Angiography Substudy. The images will be processed using a validated quantitative coronary angiography (QCA) Bifurcation software to assess quantitative data describing bifurcation geometry before and after LMCA PCI. In the Quantitative Angiography Substudy, on exploratory bases, FFRangio data reconstructed by angiographic software will be tested against stenosis LMCA lesion severity and LMCA PCI result.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with a diagnosis of documented silent ischemia, stable angina, or acute coronary syndrome (ACS).
* PCI with single or multiple drug-eluting stent (DES) for the treatment of lesion located at LMCA bifurcation and defined as a diameter stenosis of ≥50% by visual estimation.

Exclusion Criteria:

* Patients who cannot give informed consent or have a life expectancy of ≤12 months;
* Pregnant or nursing mothers. Women of child-bearing age will be asked if they are pregnant or think that they may be pregnant.
* Contraindication or suspected intolerance to anticoagulant (heparin, bivalirudin) or oral antiplatelet therapy (aspirin, clopidogrel, prasugrel, ticagrelor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of documented silent ischemia, stable angina, or ACS, undergoing PCI with single or multiple DES for the treatment of lesion located at LM coronary bifurcation and defined as a diameter stenosis of ≥50% by visual estimation.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 12 months
  The composite of: death from any cause, myocardial infarction (MI), stent thrombosis (ST), defined as definite, probable or possible following the Academic Research Consortium.

SECONDARY OUTCOMES:
Death | 12 months
  All-cause death and cardiovascular death
MI | 12 months
  Myocardial Infarction
ST | 12 months
  Stent thrombosis (definite, probable or possible)
In-hospital MACE | 12 Months
  Composite of death, MI and ST
Target Vessel Revascularization (TVR) | 12 Months
  Target Vessel Revascularization
Bleeding | 12 Months
  The occurrence of major bleeding, as a bleeding defined by the academic research consortium (BARC)- classified as type 3 (a, b or c) or 5 bleeding event

CONTACTS AND LOCATIONS:
Overall Officials: Marco Zimarino, MD, PhD, Principal Investigator — Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti

IPD SHARING:
Plan to Share IPD: Yes
Case Report Forms (CRF) will be shared among partecipating centers
Supporting Information: CSR
Time Frame: 12 Months

REFERENCES:
- [Background] Zimarino M, Briguori C, Amat-Santos IJ, Radico F, Barbato E, Chieffo A, Cirillo P, Costa RA, Erglis A, Gamra H, Gil RJ, Kanic V, Kedev SA, Maddestra N, Nakamura S, Pellicano M, Petrov I, Strozzi M, Tesorio T, Vukcevic V, De Caterina R, Stankovic G; EuroBifurcation Club. Mid-term outcomes after percutaneous interventions in coronary bifurcations. Int J Cardiol. 2019 May 15;283:78-83. doi: 10.1016/j.ijcard.2018.11.139. Epub 2018 Dec 2. PMID 30528620
- [Background] Lassen JF, Holm NR, Banning A, Burzotta F, Lefevre T, Chieffo A, Hildick-Smith D, Louvard Y, Stankovic G. Percutaneous coronary intervention for coronary bifurcation disease: 11th consensus document from the European Bifurcation Club. EuroIntervention. 2016 May 17;12(1):38-46. doi: 10.4244/EIJV12I1A7. PMID 27173860
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437